CLINICAL TRIAL: NCT03012009
Title: A Randomized Controlled Trial of a Full and a Fractional Ablative Carbon Dioxide Laser as Pretreatment for Photodynamic Therapy in the Management of Superficial Non Melanoma Skin Cancer
Brief Title: Laser Assisted Drug Delivery in the Treatment of Superficial Non Melanoma Skin Cancer: a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC/2014/0735
Record Dates: First submitted 2016-11-21; First posted 2017-01-06 (Estimated); Last update posted 2018-01-25 (Actual); Status verified 2018-01

CONDITIONS: Bowen's Disease; Superficial Basal Cell Carcinoma
Keywords: Bowen's Disease; Superficial Basal Cel Carcinoma; Non melanoma skin cancer; Photodynamic therapy; PDT; CO2 laser; Laser assisted drug delivery; Carbon dioxide laser; Laser assisted photodynamic therapy
MeSH Terms: conditions — Bowen's Disease | interventions — methyl 5-aminolevulinate; Lidocaine; Epinephrine; Anesthesia, Local

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Full ablative CO2 laser + MAL PDT (Active Comparator): The treatment starts with a full ablative CO2 laser pretreatment under local anaesthesia with injectable lidocaine hydrochloride 2% with epinephrine. This ablation is followed by photodynamic therapy: MAL is topically applied, followed by a 3 hours incubation under occlusion, whereafter 10 minutes of illumination with a LED lamp. This treatment is repeated after 14 days.
  Interventions: Device: full ablative CO2 laser; Drug: MAL; Device: LED lamp; Drug: lidocaine hydrochloride 2% with epinephrine
- Fractional ablative CO2 laser+ MAL PDT (Active Comparator): The treatment starts with a fractional ablative CO2 laser ablation under local anaesthesia with injectable lidocaine hydrochloride 2% with epinephrine. This ablation is followed by photodynamic therapy: MAL is topically applied, followed by a 3 hours incubation under occlusion, whereafter 10 minutes of illumination with LED lamp. This treatment is repeated after 14 days.
  Interventions: Device: fractional ablative CO2 laser; Drug: MAL; Device: LED lamp; Drug: lidocaine hydrochloride 2% with epinephrine

INTERVENTIONS:
Device: full ablative CO2 laser — ablation to the level of de dermal papilla
  Other Names: full ablative carbon dioxide laser
  Arms: Full ablative CO2 laser + MAL PDT
Device: fractional ablative CO2 laser — 180 micron HP, pulse 8ms, 15% overlay, 30 W (943J/cm)
  Other Names: fractional ablative carbon dioxide laser
  Arms: Fractional ablative CO2 laser+ MAL PDT
Drug: MAL
  Other Names: methyl aminolevulinate; Metvix® (Galderma)
Device: LED lamp — peak wavelength 630 nm, 37J/cm2
  Other Names: Aktilite® (Galderma); light-emitting diodes
Drug: lidocaine hydrochloride 2% with epinephrine
  Other Names: local anaesthetic; xylocaine® 2% with epinephrine

SUMMARY:
Photodynamic therapy (PDT) is a well established treatment option for superficial non melanoma skin cancer, such as superficial basal cell carcinoma (sBCC) and Bowen Disease (BD). However, a limited uptake of the topically applied photosensitizer methyl aminolevulinate (MAL) may reduce its efficacy. Pretreatment with an ablative carbon dioxide (CO2) laser has recently been studied in order to enhance the skin penetration of this photosensitizer. This study compares the results of a full ablative and a fractional ablative CO2 laser mode as pretreatment of PDT in the management of sBCC and BD. The endpoints efficacy, pain, aesthetics and patient preference are investigated during twelve months of follow up.

DETAILED DESCRIPTION:
Superficial Basal Cell Carcinoma (sBCC) and Bowen Disease (BD) are malignant skin tumors localised in the superficial epidermis. These tumors are highly prevalent in the caucasian population. Diagnosis of sBCC and BD is often delayed because the clinical manifestation may be discrete and lesions are sometimes wrongly diagnosed and treated as eczema. Once the diagnosis is established, the lesions may cover an extensive area, making surgical excision more difficult. At that moment, the physician can make use of less invasive techniques such as photodynamic therapy (PDT). Pretreatment with an ablative carbon dioxide (CO2) laser has recently been studied in order to enhance the skin penetration of the photosensitizer methyl aminolevulinate (MAL). This study compares the results of a full ablative and a fractional ablative CO2 laser mode as pretreatment of PDT in the management of sBCC and BD. Ablation of the upper epiderm of the cancer results in an deeper penetration of MAL. Fractional ablation is known to result in better wound healing compared to full ablative CO2 laser ablation, because only small skin columns are ablated instead of the entire epidermal layer. Patients with non operable sBCC or BD lesions covering an area of at least 5 cm2 or with the presence of two small separated lesions, will be investigated. Lesions greater than 5 cm2 are divided in two. After randomization, the half of the lesions will be pretreated with the full ablative CO2 laser, while the other half with the fractional ablative CO2 laser. Afterwards, the entire surface is treated with MAL-PDT. Such as in our current clinical practice, this treatment modality is repeated after a two week interval. Thus, every subject undergoes both treatment modalities, making within-patient comparison possible. The endpoints efficacy, pain, aesthetics and patient preference are investigated during twelve months of follow up.

ELIGIBILITY:
Inclusion Criteria: patients with the presence of

* non operable superficial Basal Cell Carcinoma or Bowen's Disease lesions
* and the presence of at least two lesions or the presence of one lesion covering an area greater than 5cm2

Exclusion Criteria: pregnancy and/or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Clinical efficacy after twelve months of follow up | month 12
  A three point scale with complete regression (CR), partial regression (PR) and no regression (NR) defined respectively as 100%, 25-99% and 0-25% regression.

SECONDARY OUTCOMES:
Clinical efficacy after six months of follow up | month 6
  A three point scale with complete regression (CR), partial regression (PR) and no regression (NR) defined respectively as 100%, 25-99% and 0-25% regression.
Clinical efficacy after three months of follow up | month 3
  A three point scale with complete regression (CR), partial regression (PR) and no regression (NR) defined respectively as 100%, 25-99% and 0-25% regression.
Histological efficacy after twelve months of follow up | month 12
Pain during the first treatment session | immediately after the first treatment session (day 1)
  The experienced pain during the treatment is scored bye the patient using a VAS scale of 100 mm.
Pain during the second treatment session | immediately after the second treatment session (day 14)
  The experienced pain during the treatment is scored by the patient using a VAS scale of 100 mm.
Side effects after the first treatment session | immediately after the first treatment session (day 1)
  The presence of following side effects is evaluated by the investigator: erythema, vesicles, pigment changes, scarring, infection and pain.
Side effects after one week of follow up, telephone survey | day 7
  The presence of following side effects is evaluated by the patient: erythema, vesicles, pigment changes, scarring, infection and pain.
Side effects before the second treatment session | before initiation of the second treatment session (day 14)
  The presence of following side effects is evaluated by the investigator: erythema, vesicles, pigment changes, scarring, infection and pain.
Side effects after the second treatment | immediately after the second treatment session (day 14)
  The presence of following side effects is evaluated by the investigator: erythema, vesicles, pigment changes, scarring, infection and pain.
Side effects after two weeks of follow up, telephone survey | day 21
  The presence of following side effects is evaluated by the patient: erythema, vesicles, pigment changes, scarring, infection and pain.
Side effects after three months follow up | month 3
  The presence of following side effects is evaluated by the investigator: erythema, vesicles, pigment changes, scarring, infection and pain.
Side effects after six months of follow up | month 6
  The presence of following side effects is evaluated by the investigator: erythema, vesicles, pigment changes, scarring, infection and pain.
Side effects after twelve months of follow up | month 12
  The presence of following side effects is evaluated by the investigator: erythema, vesicles, pigment changes, scarring, infection and pain.
Aesthetic result after three months of follow up | month 3
  The aesthetic result is scored by a blinded investigator using a four point scale: excellent (no significant changes), good (minor changes), poor (serious dyspigmentation, visible scarring), very poor (important scarring).
Aesthetic result after six months of follow up | month 6
  The aesthetic result is scored a by blinded investigator using a four point scale: excellent (no significant changes), good (minor changes), poor (serious dyspigmentation, visible scarring), very poor (important scarring).
Aesthetic result after twelve months of follow up | month 12
  The aesthetic result is scored a by blinded investigator using a four point scale: excellent (no significant changes), good (minor changes), poor (serious dyspigmentation, visible scarring), very poor (important scarring).
Aesthetic result according to the patient after three months of follow up | month 3
  The aesthetic result is scored by the patient using a four point scale: excellent (no significant changes), good (minor changes), poor (serious dyspigmentation, visible scarring), very poor (important scarring).
Aesthetic result according to the patient after six months of follow up | month 6
  The aesthetic result is scored by the patient using a four point scale: excellent (no significant changes), good (minor changes), poor (serious dyspigmentation, visible scarring), very poor (important scarring).
Aesthetic result according to the patient after twelve months of follow up | month 12
  The aesthetic result is scored by the patient using a four point scale: excellent (no significant changes), good (minor changes), poor (serious dyspigmentation, visible scarring), very poor (important scarring).
Technique of preference according to the patient | month 12
  Patients are asked for their preferred therapy. Following options exist: (1) full ablative CO2 laser + PDT, (2) fractional ablative CO2 laser + PDT, (3) no preference

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Boone, MD PhD, Principal Investigator — Ghent University, Dpt. of Dermatology
Locations (1):
- Department of Dermatology, Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: Undecided